CLINICAL TRIAL: NCT02869828
Title: Central Temperature Monitoring by Zero-heath-flux a Non-invasive Technic Compared to Two Invasive Technic During Surgery
Acronym: TEMP CORE BLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TEMPCORE-BLOC
Record Dates: First submitted 2016-06-20; First posted 2016-08-17 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2016-06

CONDITIONS: Major Surgery in Adult Patients

ARMS (2):
- monitoring by arterial catheter and Spot-on (Other)
  Interventions: Device: Monitoring by arterial catheter and Spot-on
- monitoring by oesophagus tube and Spot-on (Other)
  Interventions: Device: Monitoring by oesophagal probe and Spot-on

INTERVENTIONS:
Device: Monitoring by arterial catheter and Spot-on
  Arms: monitoring by arterial catheter and Spot-on
Device: Monitoring by oesophagal probe and Spot-on
  Arms: monitoring by oesophagus tube and Spot-on

SUMMARY:
Core temperature monitoring is mandatory during major surgery. The accurate techniques currently used are invasive, such as artery catheter and oesophagal probe. A new non-invasive cutaneous device, 3M SpotOn, using Zero Heath-Flux method, continuously measure core temperature. This prospective study compare the accuracy of Zero-Heath-Flux to oesophagal temperature (30 patients) and to artery catheter (20 patients) in adult patients during surgery.

DETAILED DESCRIPTION:
Every patients undergoing heavy surgery had their central temperature monitoring, through an arterial catheter if the surgery required it (30 patients in this arm), otherwise the investigators used an oesophagus tube (20 patients). We also monitored every 50 patients with a non-invasive method 3M spot on (Zero-heath-flux technic) in order to measure its fiability and validity during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo general anaesthesia for gut surgery lasting more than 2 hours
* Patients with core temperature monitored with oesophagal probe only (30 patients) or with oesophagal probe and PICCO device (20 patients)
* Patients without opposition to this study after informations given

Exclusion Criteria:

* Patients with frontal cutaneous decay wich avoid using 3M Spot-on
* Patients whom oesophagal probe was prohibited (oesophagal varices, oesophagal surgery)
* Pregnant women or breast-feeding, women who may become pregnant unless adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
temperature monitoring with Zero-Heath-Flux (SpotOn) | 1 day
temperature monitoring with oesophagal probe (Coviden) | 1 day
temperature monitoring with arterial catheter (PICCO) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- BOISSON Matthieu, Poitiers, France

REFERENCES:
- [Derived] Boisson M, Alaux A, Kerforne T, Mimoz O, Debaene B, Dahyot-Fizelier C, Frasca D. Intra-operative cutaneous temperature monitoring with zero-heat-flux technique (3M SpotOn) in comparison with oesophageal and arterial temperature: A prospective observational study. Eur J Anaesthesiol. 2018 Nov;35(11):825-830. doi: 10.1097/EJA.0000000000000822. PMID 29708906